CLINICAL TRIAL: NCT05832242
Title: Developing a Decision Tool for Diverticulitis in the Emergency Department Using Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0649
Record Dates: First submitted 2023-03-15; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simple Diverticulitis: Computed tomograpy scan showing isolated inflammation
  Interventions: Other: Ultrasound
- Complicated Diverticulitis: Computed tomograpy scan evidence of diverticulitis with either an associated abscess, fistula, obstruction, bleeding, phlegmon or perforation.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Point-of-care ultrasound in the emergency department

SUMMARY:
The purpose of this study is to create a decision tool using ultrasound, patient history, and laboratory values to predict a diagnosis of complicated diverticulitis and whether the patient requires further imaging. The accuracy of the decision tool will be evaluated. This study will also assess the ability of ultrasound to diagnose complicated and simple diverticulitis, and the inter-provider reliability of ultrasound interpretation of diverticulitis

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* Provider suspicion of diverticulitis
* CT scan ordered

Exclusion Criteria:

* Pregnant patient
* Prisoner
* Non-English speaking
* Inability to provide informed consent
* Hemodynamically unstable as determined by provider
* Previous abdominal surgery within last 7 days
* Unable to lay flat for ultrasound exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult emergency department patients suspected of having diverticulitis.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Simple Diverticulitis | 48 hours
  Computed tomography scan showing isolated inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Allison Cohen, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided